CLINICAL TRIAL: NCT04983277
Title: Study of Diabetes Mellitus and Its Complications and the Risk of Cardiovascular and Cerebrovascular Diseases
Brief Title: Diabetes Complications and the Risk of Cardiovascular and Cerebrovascular Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: DCRCCD
Record Dates: First submitted 2021-07-11; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Complications; Cardiovascular Diseases; Cerebrovascular Disease
MeSH Terms: conditions — Diabetes Complications; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes: patients with diagnosed Diabetes Mellitus
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study is intended to include 3000 diabetic patients in our hospital to collect complete medical history data, comprehensively improve the screening of diabetic complications and cardiovascular and cerebrovascular risk assessment.

DETAILED DESCRIPTION:
With the economic development and lifestyle change, the incidence and prevalence of diabetes are increasing year by year in both China and the world. Diabetics are associated with a significantly increased risk of cardiovascular and cerebrovascular disease.

It is a cross-sectional study. This study intended to include about 3000 adult patients with previously diagnosed diabetes mellitus, then collect their anthropometric data (age, gender, weight, height, waist circumference, hip circumference and etc.), life history (diet, exercise, smoking, drinking and etc.), medical history, familial medical history, clinical testing results about their diabetes complication, and make a comprehensive assessment of their cardiovascular and cerebrovascular risks. These data will be used to make further research about the diabetes complication and cardiovascular and cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic symptoms with: plasma glucose level at any time ≥11.1mmol/ L (200mg/ dL), or Fasting plasma glucose level ≥7.0mmol/ L (126mg/ dL), or plasma glucose level ≥11.1mmol/ L (200ng/ dL) for 2 h in OGTT test, or HbA1c ≥6.5%; Or those without typical symptoms should repeated the tests in another day.
* Han Chinese.
* Willingness to participate.

Exclusion Criteria:

* Secondary diabetes.
* Participants in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Framingham Risk Scose | 1 week
  The Framingham risk score calculates an individual's risk of coronary heart disease over the next 10 years based on cholesterol levels and non-cholesterol factors. Non-cholesterol factors are subdivided into risk factors, major risk factors, and other factors.
  Risk factors include: diabetes; evidence of coronary heart disease; evidence of atherosclerosis outside the heart. Major risk factors include: male older than 45 years old, female older than 55 years old; Smoking; Hypertension (higehr than 140/90mmHg or being treated for hypertension); High-density lipoprotein lower than 40 mg/dl; First-degree relatives, male younger than 55 years old, or female younger than 65 years old, with a history of coronary heart disease.
  A higher score corresponds to a higher 10-year risk of developing cardiovascular disease.
UK Prospective Diabetes Study risk score | 1 week
  This scale provides an estimate of the risks for a new coronary heart disease(CHD) event and stroke (fatal and nonfatal). The data used to calculate the UK Prospective Diabetes Study(UKPDS) risk scores (available at http://www.dtu.ox.ac.uk/riskengine/download.php) included HbA1c, systolic blood pressure, serum total cholesterol and HDL-C, atrial fibrillation, sex, age, ethnicity, smoking status, and diabetes duration. The risks of CHD, fatal CHD, stroke, and fatal stroke were estimated for 10 years.
  A higher score corresponds to a higher 10-year risk of developing cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Pengfei Shan, MD, PhD, Principal Investigator — Department of Endocrinology and Metabolism, Second Affiliated Hospital of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No